CLINICAL TRIAL: NCT05681572
Title: " Effect of Sedative and Anxiolytic Premedication on Children Experience After General Anesthesia " The pediaPREM Study.
Brief Title: Effect of Sedative and Anxiolytic Premedication on Children Experience After General Anesthesia
Acronym: pediaPREM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECHMPL21_0354; 2022-501124-23-00 (Other: EU CT (European Regulation No. 536/2014))
Record Dates: First submitted 2022-12-12; First posted 2023-01-12 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia
Keywords: children premedication; anesthesia; children perioperative experience; anxiety; sedation
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients are randomized to 2 groups to received pharmacologic premedication or placebo.
  For the premedication group, children are randomly allocated to be premedicated with either with the midazolam or dexmedetomidine (2 sup-groups).
Who Masked: Participant, Investigator
Masking Description: Physicians, the nurse responsible for administration, the staff following the patient and the patient will be blinded to randomisation.
  Only the nurse involved in the preparation of experimental treatments is not blinded. She will not be involved in the follow-up of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Premedication Group (Midazolam) (Experimental): Midazolam (0,5 mg/kg; max 10 mg), oral administration, 45 minutes prior entering in the operating room
  Interventions: Drug: Midazolam
- Premedication Group (Dexmedetomidine) (Experimental): Dexmedetomidine (2 µg/kg), oral administration, 45 minutes prior entering in the operating room
  Interventions: Drug: Dexmedetomidine
- Placebo Group (Placebo Comparator): grenadine syrup (3 mL), oral administration, 45 minutes prior entering in the operating room
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midazolam — 45 minutes before entering the operating room, patient receives the oral treatment according to their randomization arm, here Midazolam , by a blinded nurse.
  Arms: Premedication Group (Midazolam)
Drug: Dexmedetomidine — 45 minutes before entering the operating room, patient receives the oral treatment according to their randomization arm, here Dexmedetomidine , by a blinded nurse.
  Arms: Premedication Group (Dexmedetomidine)
Drug: Placebo — 45 minutes before entering the operating room, patient receives the oral treatment according to their randomization arm, here Grenadine Syrup, by a blinded nurse.
  Arms: Placebo Group

SUMMARY:
Children undergoing general anesthesia for surgery commonly need sedative and anxiolytic premedication but little clinical evidence supports is benefit for children older than 7 years old.

The aim of this prospective randomized clinical trial is to assess the impact of pharmacologic premedication on perioperative children experience.

DETAILED DESCRIPTION:
Surgery is a stressful experience in children with preoperative and postoperative anxiety.

For preschooler undergoing surgery, anxiety is the highest in the preoperative period.

Most of studies have been conducted on young children (< 7yrs old) to show the relationship between preoperative anxiety and emergence of delirium and postoperative maladaptive behavioral changes.

Sedative and anxiolytic medication is frequently used in children to reduce anxiety and postoperative maladaptive experiences. Nevertheless, little clinical evidence supports is benefit for children older than 7 years.

Treating anxiety is not necessarily associated with better experience in all children because premedication causes postoperative sedation, amnesia and cognitive impairment.

The aim of this prospective randomized clinical trial is to assess the impact of pharmacologic premedication on perioperative children experience using self-report questionnaire.

Patients are randomized to 2 groups to received pharmacologic premedication or placebo.

For the premedication group, children are randomly allocated to be premedicated with either with the midazolam or dexmedetomidine

ELIGIBILITY:
Inclusion Criteria:

* Subject over 7 and under 18 years of age
* Subjects who are scheduled for surgery
* Subject who will be under general anesthesia
* Subject able to complete a self-questionnaire in French

Exclusion Criteria:

* Subject who has already participated in the pediaPREM study
* Subject with a treated anxiety disorder
* Subject with cognitive disorders
* Subject suffering from chronic pain (outside the operated area)
* Subject with ADD (Attention Deficit Disorder) with or without hyperactivity, with or without treatment
* Subject suffering from mental retardation
* Subjects receiving psychotropic treatment
* Subject whose intervention could reduce the ability to complete a self-questionnaire (neurosurgery etc.)
* Subject with a contra-indication to midazolam and its excipients
* Subject with a contra-indication to dexmedetomidine and its excipients
* Subjects who need to receive intravenous alpha agonist in perioperative
* Subjects requiring emergency intervention
* Subjects requiring preoperative hypnosis
* Subject who needs general anesthesia for diagnostic purposes (biopsy, etc...)
* Subject having had a surgical intervention in the month preceding the inclusion.
* Subject who will have an iterative surgical intervention within 15 days (removal of material, burns etc...)
* Subjects who are scheduled for surgery as part of oncology management
* Pregnant or breastfeeding woman
* Subject whose two parents have not signed a written informed consent
* Subjects who are not affiliated with or benefiting from a social security plan

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2027-10-18 (Estimated)

PRIMARY OUTCOMES:
EVANpedia Score | from the day of surgery up to the day one after surgery
  To evaluate patient experience of the perioperative and post-operative period

SECONDARY OUTCOMES:
VAS-anxiety Scores | from preoperative period up to 6 postoperative month
  To evaluate the perioperative level of anxiety thanks to the Visual Analogue Scale (VAS)
Postoperative waking delay | from the end of the surgery up to the exit of the recovery room
  Time to wake up after surgery (minutes) to evaluate the delay emergence from anesthesia
Modified Brice questionnaire Score | from the day of surgery up to 1 day
  To evaluate postoperative amnesia after anesthesia
Post Hospitalization Behavior Scores | 15 postoperative days
  To evaluate changes of behavioral (appetite, sleep, sociability) after surgery
quality of life | 6 postoperative months
  to evaluate the impact of the perioperative experience on the long-term experience
neuropathic pain | 6 postoperative month
  to evaluate the percentage of patients with long-term neuropathic pain
FPS-r scores | from the end of the surgery up to 6 post-operative month
  To evaluate the Postoperative level of pain thanks to the Faces Pain Scale-revised (FPS-r)
Quality of life PedsQL | Up to 6 months post-operatively
  The quality of life will be measured by PedsQL in order to evaluate the impact of the perioperative experience on the long-term experience. The 23 questions cover 4 different domains: physical functioning (8 items), emotional functioning (5 items), social functioning (5 items) and academic functioning (5 items).
  The parent questionnaire assesses parents' perceptions of their child's health-related quality of life. On the PedsQL Generic Core Scales, for ease of interpretability, items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DADURE, PHD, Study Director — Hospital of Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France